CLINICAL TRIAL: NCT03521401
Title: Effects of Exercise on Young Adult Women With ACEs: an Integrative Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ED17157; P20GM109097 (NIH)
Record Dates: First submitted 2018-03-29; First posted 2018-05-11 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Life Experiences
Keywords: Adverse Childhood Experiences; Exercise Intervention; Inflammation; Resilience; Health
MeSH Terms: conditions — Inflammation | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ACE - Exercise Group (Experimental): Participants with ACE scores of 4 or higher who will undergo exercise training for the duration of the study (experimental).
  Interventions: Behavioral: Exercise
- ACE - Non-Exercise Group (No Intervention): Participants with ACE scores of 4 or higher who will not undergo exercise training for the duration of the study (+ control).
- Non-ACE - Non-Exercise Group (No Intervention): Participants with ACE scores of 0 who will not undergo exercise training for the duration of the study (- control).

INTERVENTIONS:
Behavioral: Exercise — Participants assigned to the exercise group will undergo structured, progressive resistance and aerobic exercise for 8 weeks. Resistance training and aerobic training will each be completed twice weekly for a total of 16 resistance and 16 aerobic exercise training sessions.
  Arms: ACE - Exercise Group

SUMMARY:
The process by which the body responds to stressors to maintain homeostasis is called allostasis and is dependent on the integrated function of the nervous, endocrine, and immune systems. ACEs adversely affect these system, cause allostatic load, and can modify development of allostatic systems. However, the central hypothesis is that exercise can reduce allostatic load by positively augmenting function of each of these three systems. No previous studies have examined the effects of structured exercise interventions in individuals with ACEs. The investigators are studying the effects of 8-weeks of structured resistance and aerobic exercise on biomarkers related to nervous, endocrine, immune, and metabolic function and several clinical outcomes in young adult women with ACEs. The specific aims will test several hypotheses, and are as follows: SPECIFIC AIM 1: Conduct a feasibility study to explore whether progressive, structured exercise can help mitigate the adverse physiological effects of stress and trauma early in life. SPECIFIC AIM 2: Determine whether progressive, structured exercise can help improve health-related quality of life, anxiety, and traits like hope, self-efficacy, or self-control, resilience. SPECIFIC AIM 3: Determine whether the type and timing of exposure to ACEs has a significant influence on the severity of psychopathology and long-term physiological response to ACEs.

ELIGIBILITY:
Inclusion Criteria:

1. provide written and dated informed consent to participate in the study;
2. be willing and able to comply with the protocol;
3. be between the ages of 18 and 29, inclusive;
4. be free from chronic cardiovascular, pulmonary, or musculoskeletal disease as determined by a health history questionnaire;
5. not currently prescribed or taking anti-inflammatory or lipid-lowering medications;
6. have either an ACE score of 0 or 4 or higher;
7. have a BMI between 18.5 and 40.0, inclusive;
8. not enrolled in another clinical trial within thirty days prior to enrollment; and
9. answer no to all questions on the PAR-Q for people aged 15 to 69, which assesses a person's eligibility to engage in exercise without contraindications.

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2019-11-10 (Actual)

PRIMARY OUTCOMES:
C-reactive protein | 8-weeks
  C-reactive protein concentrations (mg/L) will be examined from blood samples taken before- and after- the 8-week training or control period.
Brain-Derived Neurotrophic Factor | 8-weeks
  Plasma concentrations of brain-derived neurotrophic factor (BDNF; pg/mL), a biomarker of neurogenesis, will be examined from blood samples taken before- and after- the 8-week training or control period.
Skeletal muscle size | 8-weeks
  Ultrasound based assessments of skeletal muscle size (cm^2) will be obtained before- and after- the 8-week training or control period.
Skeletal muscle strength | 8-weeks
  Skeletal muscle strength (Newton meters [Nm]) will be determined before- and after- the 8-week training or control period.
TNF-alpha | 8-weeks
  TNF-alpha concentrations (pg/mL) will be examined from blood samples taken before- and after- the 8-week training or control period. TNF-alpha is a cytokine involved in systemic inflammation.
Interleukin-1 receptor agonist | 8-weeks
  Interleukin-1 receptor agonist concentrations (pg/mL) will be examined from blood samples taken before- and after- the 8-week training or control period.
Skeletal muscle function | 8-weeks
  Motor unit behavior will be assessed utilizing surface electromyographic signal decomposition, which will be collected while participants perform submaximal isometric (i.e., static) muscle actions. These signals will be collected before- and after- the 8-week training or control period. To examine motor unit behavior, the relationship between motor unit recruitment threshold versus firing rate will be determined for all detected motor units for an individual subject.
Cortisol | 8-weeks
  Concentrations of salivary cortisol (µg/dL), a stress hormone, will be obtained twice in one day (8 h between samples) before- and after- the 8-week training or control period.

SECONDARY OUTCOMES:
Health-related quality of life | 8-weeks
  Health-Related Quality of Life: The RAND 36-item short form survey instrument (SF-36) will be used to assess health-related quality of life (HQROL) before- and after- the 8-week training or control period. This will serve as an overall assessment of each individuals' perception of their health.
Anxiety | 8-weeks
  Participants' levels of anxiety will be assessed using the Zung Self-Rating Anxiety Scale (SAS) before- and after- the 8-week training or control period.
Depression | 8-weeks
  Participants' levels of depression will be measured utilizing the Center for Epidemiologic Studies Depression Scale Revised (CESD-R) before- and after- the 8-week training or control period.
Resiliency | 8-weeks
  Participants' resiliency will be measured using the Connor-Davidson Resilience Scale before- and after- the 8-week training or control period.
Hope | 8-weeks
  Participants' levels of hope will be assessed with the 12-item adult hope scale before- and after- the 8-week training or control period.
Monocyte Heterogeneity | 8-weeks
  The heterogeneity of monocyte populations will be determined from the white blood cells in blood plasma using flow cytometry. The relative number (%) of CD14++CD16- vs. CD14+CD16++ vs. CD14++CD16+ monocytes will be determined for each participant before- and after- the 8-week training or control period.

OTHER OUTCOMES:
Fasting glucose concentrations | 8-weeks
  Fasting blood glucose concentrations (mg/dL) will be determined for each participant before-, during (week 4), and after- the 8-week training or control period.
Fasting lipid concentrations | 8-weeks
  Fasting blood lipid concentrations (mg/dL) will be determined for each participant before-, during (week 4), and after- the 8-week training or control period.
Fasting choleterol concentrations | 8-weeks
  Fasting blood cholesterol concentrations (mg/dL) will be determined for each participant before-, during (week 4), and after- the 8-week training or control period.
Self Efficacy | 8-weeks
  Participants' levels of self-efficacy will be assessed with the General Self-Efficacy Scale before- and after- the 8-week training or control period.
Self Esteem | 8-weeks
  Participants' levels of self-efficacy will be assessed with the Rosenberg Self-Esteem Scale before- and after- the 8-week training or control period.
Grit | 8-weeks
  Participants' levels of Grit will be measured using the 12-item Grit scale, which assesses passion and perseverance for achieving long-term goals, before- and after- the 8-week training or control period.

CONTACTS AND LOCATIONS:
Locations (1):
- 192 Colvin Recreation Center, Stillwater, Oklahoma, United States